CLINICAL TRIAL: NCT00441987
Title: A Single Ascending Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GSI-953 Administered Orally to Healthy Japanese Male Subjects and Healthy Elderly Male Japanese Subjects.
Brief Title: Study Evaluating the Safety and Pharmacokinetics of a Single Dose of GSI-953
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3183A1-101
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2022-05-03 (Actual); Status verified 2010-06

CONDITIONS: Healthy
Keywords: Japanese; Healthy; Alzheimers Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- Single Dose of GSI-953 (Experimental)
  Interventions: Drug: GSI-953

INTERVENTIONS:
Drug: GSI-953

SUMMARY:
The purpose of the protocol is to assess the initial pharmacokinetic (PK) profile of a single oral dose of GSI-953 to healthy male Japanese subjects and healthy elderly male Japanese subjects.

ELIGIBILITY:
* Healthy males aged 20 - 40 and healthy males aged greater than 65.
* Body mass index range of 17.6 - 26.4 kg/m2 greater than or equal to 45 kg.
* Non-smokers or smoker of fewer than 10 cigarettes a day.

Ages: 20 Years to 120 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2007-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting Adverse Event | 10 months
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Kitashinagawa, Shinagawa-ku, Japan